CLINICAL TRIAL: NCT01596634
Title: A Pilot Study of Bovine Lactoferrin in Patients With Colorectal Carcinoma Receiving Oxaliplatin-Based Chemotherapy and Self-Reported Taste Disturbances
Brief Title: Bovine Lactoferrin in Reducing Taste Disturbances in Patients With Colorectal Cancer Receiving Oxaliplatin-Based Chemotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00020136; NCI-2012-00279 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CCCWFU 98112 (Other: Wake Forest University Health Sciences)
Record Dates: First submitted 2012-05-09; First posted 2012-05-11 (Estimated); Last update posted 2018-07-03 (Actual); Status verified 2018-07

CONDITIONS: Colorectal Cancer; Dysgeusia; Oral Complications of Chemotherapy
MeSH Terms: conditions — Colorectal Neoplasms; Dysgeusia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supportive care (bovine lactoferrin) (Experimental): Patients receive bovine lactoferrin PO (rinse or tablet) TID for 1 month. Treatment continues in the absence of unacceptable toxicity.
  Interventions: Other: questionnaire administration; Procedure: quality-of-life assessment; Other: laboratory biomarker analysis; Dietary Supplement: bovine lactoferrin

INTERVENTIONS:
Other: questionnaire administration — Ancillary studies
Procedure: quality-of-life assessment — Ancillary studies
  Other Names: quality of life assessment
Other: laboratory biomarker analysis — Correlative studies
Dietary Supplement: bovine lactoferrin — Given PO

SUMMARY:
The purpose of this research study is to determine if using a lactoferrin supplement will improve taste perception. Lactoferrin is a type of protein that is naturally produced in the body and is commonly found in saliva.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the impact of lactoferrin (bovine lactoferrin) supplementation on self-reported taste and smell disturbances in patients with colorectal cancer receiving oxaliplatin-based chemotherapy

SECONDARY OBJECTIVES:

I. To assess the impact of lactoferrin supplementation on the baseline lipid peroxidation byproducts in saliva in these patients as measured by the thiobarbituric acid-reactive substances (TBARs) assay.

II. To assess the impact of lactoferrin supplementation on the ability of these patients to generate increased lipid peroxidation byproducts when challenged with a weak iron containing solution.

III. To assess the impact of lactoferrin supplementation on self-reported general quality of life and on specific self-reported anorexia/cachexia issues in patients with established chemotherapy-induced taste disturbances.

IV. To assess the incidence of vitamin D deficiency in patients with oxaliplatin-based therapy induced taste changes

OUTLINE:

Patients receive bovine lactoferrin orally (PO) (rinse or tablet) thrice daily (TID) for 1 month. Treatment continues in the absence of unacceptable toxicity.

After completion of study treatment, patients are followed up at 2 and 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed colorectal carcinoma
* There are no restrictions on the amount or types of prior therapy
* Eligible patients must be receiving ongoing chemotherapy with an oxaliplatin containing-regimen which is planned to continue for at least one month following enrollment in this trial
* Any dose or schedule of oxaliplatin administration is allowed as long as patients have self-reported taste disturbance that has either:

  * 1) developed since the initiation of oxaliplatin-based therapy, or
  * 2) a pre-existing, treatment-induced taste disturbance has subjectively worsened since initiating oxaliplatin-based therapy
* Patients must have normal baseline self-reported taste perception prior to the development of colorectal carcinoma
* Life expectancy of >= 3 months
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients with a subjective history of an extreme dry mouth syndrome that prevents them from producing adequate amounts of saliva (approximately 2 mL in 15-20 min)
* Patients known to be human immunodeficiency virus (HIV)-positive
* Patients with any of the following conditions: untreated gastrointestinal reflux disease; untreated diabetes mellitus; active thrush; active oral infection; active mucositis
* Patients who are known to be pregnant or who are breastfeeding are excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2015-08 (Actual); Study Completion 2015-10-10 (Actual)

PRIMARY OUTCOMES:
Change in the Taste Visual Analog Scale (VAS) and taste and smell questionnaire responses | Approximately 1 month
  Paired-tests will be used to assess the significance of these changes. Linear regression models will be used to determine which patient covariates are associated with change. Repeated measures models will also be used to assess the changes over time using all the repeated measures and contrasts will be used to assess individual pair-wise differences. Descriptive reports will consist of summary statistics (means, standard deviations, proportions, etc.).

SECONDARY OUTCOMES:
Effect of bovine lactoferrin on lipid peroxidation byproducts in saliva as measured by the TBARs assay | Approximately 2 months
Malondialdehyde (MDA) concentrations before and after a ferrous iron oral rinse | Approximately 2 months
Quality of life as quantified by the Functional Assessment of Anorexia/Cachexia Treatment (FAACT) questionnaire | Approximately 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Lesser, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Comprehensive Cancer Center of Wake Forest University, Winston-Salem, North Carolina, United States